CLINICAL TRIAL: NCT04368832
Title: ImPROving prenaTal carE During ConfinemenT: Impact of Confinement on the Quality of Prenatal Care Perceived in Low-risk Pregnancy
Brief Title: imPROving prenaTal carE During ConfinemenT
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mme Gaëlle AMBROISE, Mrs, Central Hospital, Nancy, France
Other Study IDs: 2020-A01023-36
Record Dates: First submitted 2020-04-22; First posted 2020-04-30 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related; COVID
Keywords: COVID-19; containment measures
MeSH Terms: conditions — COVID-19 | interventions — Remote Consultation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: During prenatal monitoring, at least one consultation by remote consultation (phone or teleconsultation)
  Interventions: Other: Remote consultation
- Control group: Prenatal monitoring by face-to-face consultations adapted to confinement (absence of clinical signs or notion of travel, occupation, contact, clustering (TOCC), no attendant, limited movements inside the hospital and precautions of "droplet" and "contact" type)

INTERVENTIONS:
Other: Remote consultation — One or more consultation is conducted by phone or teleconsultation during prenatal monitoring
  Groups: Experimental group

SUMMARY:
This study is a non-randomized, quasi-experimental, monocentric study comparing two prenatal monitoring modes in low-risk pregnancy: including at least one remote consultation (phone or teleconsultation) versus face-to-face adapted to confinement. The quality of care perceived by the pregnant women were evaluated according to monitoring modes set up during the COVID-19 pandemic confinement period. The women included planned to give birth at the regional academic Maternity of Nancy, France.

DETAILED DESCRIPTION:
The emergency confinement measures deployed by most industrialized countries governments to limit the impact of the coronavirus disease 2019(COVID-19) pandemic resulted in rapid and unpredictable changes in methods of obstetric monitoring. International and French government recommendations called for a reorganization of mandatory monitoring, particularly for low-risk pregnancies (limit the presence of the coparent during follow-up consultations and implement remote consultations). The potential impact of this reorganization on care perception, probably increased by the context of an unprecedented economic, social and health crisis, is unpredictable. In the absence of a previous event of comparable importance, it is impossible to anticipate differences in satisfaction with antenatal management and in stress level between women exposed to the two types of monitoring. Many factors can influence the perception of care quality, such as the socio-economic environment and the level of health literacy, that is, the individual's ability to find information on health, to understand and use this information to improve his own health or develop autonomy in health care system.

The objective of this study is to determine which type of monitoring is better perceived by pregnant women, the factors associated with this perception and the links with the level of knowledge and mastery of women regarding reproductive health and digital tools.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman eligible for type A or A1 follow-up according to the French Health Authority "Haute Autorité de Santé" (HAS) (low-risk pregnancy)
* Having consulted at least one practitioner (midwife or physician) during the COVID-19 national confinement period
* Gestational age > 7 weeks of amenorrhea on 17th March 2020, at the beginning of the national confinement period in France
* having received complete information on the organisation of this research and not opposed to participation and exploitation of her data
* Childbirth expected in the regional academic Maternity of Nancy
* Member of or beneficiary of a social security scheme
* Speaking French and able to complete a self questionnaire or having the possibility of being assisted

Exclusion Criteria:

* Not understanding French
* Multiple pregnancy
* Request for voluntary termination of pregnancy
* Discovery or suspicion of congenital malformation
* Under protection of justice, guardianship or trusteeship
* Deprived of liberty by judicial or administrative decision
* Undergoing psychiatric care under sections L. 3212-1 and L. 3213-1 of french law (hospitalization without consent).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women with low obstetrical risk expecting to give birth in the Maternité régionale universitaire de Nancy, France.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Score of perceived quality of prenatal care | Through study completion, an average of 3 months, ie either at the beginning of the second or the third trimester of pregnancy, or during immediate postpartum care
  score obtained with the Quality of prenatal care questionnaire (QPCQ) as close as possible after release from containment

SECONDARY OUTCOMES:
Level of stress during pregnancy | Through study completion, an average of 3 months, ie at the beginning of the second and the third trimester of pregnancy, and during immediate postpartum care
  Perceived stress measured with Perceived Stress Scale-10 (PSS-10) scale
level of health and digital literacy | Through study completion, an average of 3 months, ie at the beginning of the second and the third trimester of pregnancy, and during immediate postpartum care
  level of health and digital literacy evaluated with Health Literacy Questionnaire (HLQ) and eHealth Literacy Questionnaire (eHLQ) questionnaire
Obstetrical outcomes | Through study completion, an average of 6 months, ie at the end of postpartum care hospitalization
  core set of outcomes for maternity care
Characteristics of medical supervision during pregnancy | Through study completion, an average of 6 months, ie throughout the period of pregnancy
  Number of remote, face-to-face or emergency consultations during pregnancy and requester of each consultation (patient or practitioner)

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle Ambroise, Principal Investigator — CHRU Nancy
Locations (1):
- Maternité Régionale Universitaire de Nancy, Nancy, France

REFERENCES:
- [Derived] Avercenc L, Ngueyon Sime W, Bertholdt C, Baumont S, Freitas AC, Morel O, Guillemin F, Ambroise Grandjean G. Improving prenatal care during lockdown: Comparing telehealth and in-person care for low-risk pregnant women in the PROTECT pilot study. J Gynecol Obstet Hum Reprod. 2022 Nov;51(9):102445. doi: 10.1016/j.jogoh.2022.102445. Epub 2022 Jul 24. PMID 35882366